CLINICAL TRIAL: NCT01749995
Title: Prospective Validation of the Use of the Freund Clock Drawing Test (CDT) to Screen for Cognitive Dysfunction in Cancer Patients Undergoing Comprehensive Geriatric Assessment (CGA)
Brief Title: Validation of the Freund Clock Drawing Test to Screen for Cognitive Dysfunction in Cancer Patients
Acronym: PROACTIVE
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Dr. Philip Debruyne, Consultant Medical Oncologist, General Hospital Groeninge
Other Study IDs: AZGS2012061
Record Dates: First submitted 2012-12-11; First posted 2012-12-17 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Elderly Cancer Patients; Cognitive Impairment
Keywords: Elderly cancer patients; Screening tool; Cognitive impairment; Freund Clock Drawing Test
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A Comprehensive Geriatric Assessment (CGA) has become a fundamental aid in the evaluation and treatment planning of older cancer patients. Systematic reviews of trials of geriatric assessments have shown effectiveness when interventions are implemented. Although CGA is a fundamental tool in the care of the geriatric patient, the integration and application of this tool in oncologic practice are still in evolution. Cognition is one of the domains examined within a CGA. Studies have noted that up to 25% to 50% of older patients had cognitive abnormalities that warranted further evaluation. Cognitive dysfunctions can influence the ability to weigh the risks and benefits of cancer therapy, to comply with the suggested treatment plan, and to recognize the symptoms of toxicity that need medical attention. Recently, the Freund Clock Drawing Test (CDT) has been proposed as a quick and simple screening tool to assess cognitive dysfunction. A retrospective analysis on 105 cancer patients at the General Hospital Groeninge showed that a cut-off score of ≤ 4 for the CDT has a good AUC, sensitivity and specificity.

Aims

1. To validate the Clock Drawing Test as a screening tool to identify elderly cancer patients in need of a more in-depth cognitive evaluation within a comprehensive geriatric assessment (CGA)
2. Further registration of data in a database coupled to the Cancer Registry in the General Hospital Groeninge as set up by the PROGERCAN study

DETAILED DESCRIPTION:
Design: A prospective, observational, cohort study. All geriatric patients who are diagnosed with cancer will be screened by an oncology clinical nurse specialist or study collaborator with the G8 questionnaire. Patients who screen positive, will be refered to the multi-disciplinary onco-geriatric program where a member of the geriatric oncology team will implement a comprehensive geriatric evaluation under supervision of an oncologist and/or geriatrician, who will then formulate recommendations and might suggest referral to other health care providers.

Population: All consenting patients, aged ≥ 70, who are referred for anti-cancer treatment in the General Hospital Groeninge and who are in need of a CGA.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have reached the age of 70 or more at the moment of enrolment
* Patients should be eligible for standard CGA as per local practice (e.g. on the basis of positive screening with G8 or referred by a treating physician on the basis of clinical suspicion of vulnerability or frailty)
* Histologically confirmed diagnosis of cancer. All stages of cancer are eligible.
* Patients should be fluent in Dutch or French
* Patients must receive their primary oncology care (surgery, course of (neo)adjuvant or palliative chemotherapy, radiotherapy, targeted therapy, palliative care, experimental treatment as part of a clinical trial,...) planned in the General Hospital Groeninge
* Patients can be included before or at the start of a line of treatment but not during a line of treatment
* Patients should have signed informed consent

Exclusion Criteria:

* Patients who do not match the inclusion criteria
* Patients who are visiting the oncology clinic for a second opinion and do not wish to be treated in the General Hospital Groeninge
* Patients who already started a respective line of treatment
* Patients deemed fit on the basis of negative screening (negative result on G8) unless the treating physician suspects vulnerability or frailty based on clinical judgement

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consenting patients, aged ≥ 70, who are referred for anti-cancer treatment in the General Hospital Groeninge and who are in need of a CGA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip R Debruyne, MD, PhD, MSc, FRCP, Principal Investigator — AZ Groeninge
Locations (1):
- General Hospital Groeninge, Cancer Center, Kortrijk, Belgium

REFERENCES:
- [Background] Ketelaars L, Pottel L, Lycke M, Goethals L, Ghekiere V, Santy L, Boterberg T, Van Den Noortgate N, Pottel H, Debruyne PR. Use of the Freund clock drawing test within the Mini-Cog as a screening tool for cognitive impairment in elderly patients with or without cancer. J Geriatr Oncol. 2013 Apr;4(2):174-82. doi: 10.1016/j.jgo.2012.10.175. Epub 2012 Nov 2. PMID 24071542
- [Result] Lycke M, Ketelaars L, Boterberg T, Pottel L, Pottel H, Vergauwe P, Goethals L, Van Eygen K, Werbrouck P, Debruyne D, Derijcke S, Borms M, Ghekiere V, Wildiers H, Debruyne PR. Validation of the Freund Clock Drawing Test as a screening tool to detect cognitive dysfunction in elderly cancer patients undergoing comprehensive geriatric assessment. Psychooncology. 2014 Oct;23(10):1172-7. doi: 10.1002/pon.3540. Epub 2014 Apr 11. PMID 24729471

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Older patients with cancer receiving a full CGA
Period: Overall Study
Arm/Group | Cohort
Started | 200
Completed | 196
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Cohort
Number analyzed (Participants) | 196
Age, Continuous [Mean (Full Range); unit: years] | 79.0 [70.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 196

OUTCOME MEASURES:

1. Primary Outcome: Validation of the Freund Clock Drawing Test, and Its Predefined Cut-off of ≤ 4, as a Screening Tool to Identify Elderly Cancer Patients in Need of a More In-depth Cognitive Evaluation With the Folstein MMSE Within Comprehensive Geriatric Assessment
Description: A Receiver Operating Characteristic (ROC) analysis was applied in order to validate the Freund Clock Drawing Test at its predefined cut-off of ≤ 4. This ROC analysis illustrates the capacity of the Freund Clock Drawing Test to identify elderly cancer patients in need of a more in-depth cognitive evaluation with the Folstein MMSE within comprehensive geriatric assessment. The ROC curve is a fundamental tool for diagnostic test evaluation. In a ROC curve the true positive rate (Sensitivity) is plotted in function of the false positive rate (100-Specificity) for different cut-off points of a parameter. The AUC (Area Under Curve) is the area enclosed by the ROC curve. The range of possible AUC values is [0, 1]. A perfect classifier has AUC = 1 and a completely random classifier has AUC = 0.5. Usually, themodel will score somewhere in between.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: unitless
Arm/Group | Cohort
Number analyzed (Participants) | 196
unitless | 0.95 [0.78 to 1.00]

2. Primary Outcome: Further Registration of Data in a Database Coupled to the Cancer Registry in the General Hospital Groeninge as Set up by the PROGERCAN Study
Description: During the PROGERCAN study, a database was set up in which the results of the CGA were coupled to the data available in the Cancer Registry of the General Hospital Groeninge. In this project, we aim continue this registration.
Time Frame: Baseline
Reporting Status: Not Posted

3. Secondary Outcome: Evaluation of the Mini-Cog (Cognitive Screening Tool Consisting of a Clock Drawing With 3-word Recall Test) When Using the Freund CDT
Time Frame: Baseline
Reporting Status: Not Posted

4. Secondary Outcome: To Determine the Time-saving
Description: Determination of the time-saving when using the Freund Clock Drawing Test instead of the Folstein MMSE
Time Frame: Baseline
Reporting Status: Not Posted

5. Secondary Outcome: To Compare the Freund Scoring System With Other Scoring Systems (Such as Watson and Colleagues), When Using a Predrawn Circle
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: To Develop a Tumour Tissue Database (Bio Bank) of Elderly Cancer Patients, Solely for Scientific Purposes
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: There were no adverse event data collected as this was an observational study.
Description: There were no risks related to participation to our trial, as this was an observational study. Therefore, no adverse event, mortality rates or risk for serious adverse event data were collected.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes